CLINICAL TRIAL: NCT05030818
Title: Cross-over Analysis of the Control of Coronary Risk Factors and Level of Platelet Inhibition With a Polypill
Brief Title: Cross-over Study of Coronary Risk Factors With a Polypill
Acronym: POLICROSS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación EPIC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: POLICROSS
Record Dates: First submitted 2021-08-30; First posted 2021-09-01 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Coronary Artery Disease
Keywords: Hypertension; LDL-cholesterol; Platelet inhibition
MeSH Terms: conditions — Coronary Artery Disease; Hypertension | interventions — Ramipril; Atorvastatin

STUDY DESIGN:
Intervention Model Description: Each patient will be treated (Randomized) during 3 months with the polypill acetylsalicylic acid, ramipril and atorvastatin) and another 3 months with the same drugs and at the same doses than the polypill
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polypill (Experimental): Patients will be receiving the polypill at the adequate doses during 3 months
  Interventions: Drug: Drugs taken separately: acetylsalicylic acid, ramipril and atorvastatin
- Drugs taken separately (Active Comparator): Patients will be receiving during 3 months the same components and at the same doses than with the polypill
  Interventions: Drug: Polypill of acetylsalicylic acid, ramipril and atorvastatin

INTERVENTIONS:
Drug: Polypill of acetylsalicylic acid, ramipril and atorvastatin — Administration of acetylsalicylic acid, ramipril and atorvastatin in a polypill during 3 months more
  Arms: Drugs taken separately
Drug: Drugs taken separately: acetylsalicylic acid, ramipril and atorvastatin — Patients will be receiving during 3 months more the same components acetylsalicylic acid, ramipril and atorvastatin than with the polypill
  Arms: Polypill

SUMMARY:
Open-label, randomized, cross-over study conducted in a single center, applied to patients receiving a polypill with 100 mg of acetyl salicylic acid and different doses of ramipril and atorvastatin for indication of secondary prevention according to clinical practice, with objective of analyzing the level of systolic blood pressure and LDL-cholesterol in the same patient in 2 different periods: one under treatment of 3 months with the polypill and another of 3 months with the components separately.

DETAILED DESCRIPTION:
The European Society of Cardiology indicates that reducing the frequency of administration is the most effective measure to improve therapeutic adherence. Current guidelines recommend with class I and level of evidence A the use of polypills.

A polypill, composed of 100 mg of acetylsalicylic acid and variable doses of atorvastatin and ramipril, is approved for secondary prevention of cardiovascular disease and has also been widely used in primary prevention.

Numerous studies have been carried out focusing on different designs of polypill in cardiovascular prevention to study their efficacy, cost-effectiveness and administration schedule. Specifically, that polypill already has an extensive literature. However, although there are previous studies with a cross-over design with other types of polypill to assess the effects on the control of arterial hypertension and LDL cholesterol, to date there has never been a cross-over design study with the polypill compared to the administration of its components separately in the control of blood pressure, lipid level and level of platelet aggregation.

Patients will be randomized to polypill vs separate components. Each patient will receive a follow-up visit per month for 6 months, of which will be 3 consecutive months with treatment with the polypill in its corresponding dose and the remaining 3 months with the same drugs separately.

Primary objectives: Systolic blood pressure level and LDL cholesterol. Secondary objectives: Degree of platelet aggregation with thromboxane A2 kit, diastolic blood pressure level, total cholesterol and HDL, level of patient satisfaction, degree of adherence to treatment, adverse events.

ELIGIBILITY:
Inclusion Criteria:

Patients over 18 years of age. Patients under treatment with the Trinomia® polypill in any of its presentations for indication of secondary prevention and who can make the 6 visits necessary to complete the study. Patients who sign the Informed Consent.

Exclusion Criteria:

Patients who do not sign the informed consent. Patients with an inability to understand and comply with the protocol. Patients with contraindication to any component of the polypill. Patients who are already participating in another clinical trial. Patients with any condition that limits life expectancy to <1 year. Patients with programmed coronary revascularization. Patients with coronary stent implantation in the last 12 months. Patients treated with any antithrombotic drug in addition to acetylsalicylic acid, that is, low molecular weight heparin, P2Y12 receptor inhibitors, or oral anticoagulants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2022-10-14 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
LDL-cholesterol | Months 2 and 3 vs. Months 5 and 6
  Mean of absolute level of LDL cholesterol
Systolic blood pressure | Months 2 and 3 vs. Months 5 and 6
  Mean of absolute level of systolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Iñigo Lozano, MD, PHD, Principal Investigator — Hospital de Cabueñes, Gijon
Locations (1):
- Hospital Universitario de Cabueñes, Gijón, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tamargo J, Castellano JM, Fuster V. The Fuster-CNIC-Ferrer Cardiovascular Polypill: a polypill for secondary cardiovascular prevention. Int J Cardiol. 2015 Dec;201 Suppl 1:S15-22. doi: 10.1016/S0167-5273(15)31028-7. PMID 26747390
- [Result] Castellano JM, Sanz G, Penalvo JL, Bansilal S, Fernandez-Ortiz A, Alvarez L, Guzman L, Linares JC, Garcia F, D'Aniello F, Arnaiz JA, Varea S, Martinez F, Lorenzatti A, Imaz I, Sanchez-Gomez LM, Roncaglioni MC, Baviera M, Smith SC Jr, Taubert K, Pocock S, Brotons C, Farkouh ME, Fuster V. A polypill strategy to improve adherence: results from the FOCUS project. J Am Coll Cardiol. 2014 Nov 18-25;64(20):2071-82. doi: 10.1016/j.jacc.2014.08.021. Epub 2014 Sep 1. PMID 25193393
- [Result] Castellano JM, Verdejo J, Ocampo S, Rios MM, Gomez-Alvarez E, Borrayo G, Ruiz E, Ibanez B, Fuster V; SORS investigators. Clinical Effectiveness of the Cardiovascular Polypill in a Real-Life Setting in Patients with Cardiovascular Risk: The SORS Study. Arch Med Res. 2019 Jan;50(1):31-40. doi: 10.1016/j.arcmed.2019.04.001. Epub 2019 Apr 19. PMID 31101241
- [Result] Gonzalez-Juanatey JR, Tamargo J, Torres F, Weisser B, Oudovenko N. Pharmacodynamic study of the cardiovascular polypill. Is there any interaction among the monocomponents? Rev Esp Cardiol (Engl Ed). 2021 Jan;74(1):51-58. doi: 10.1016/j.rec.2019.11.008. Epub 2020 Jan 23. English, Spanish. PMID 31983653
- [Result] Marzal D, Rodriguez Padial L, Arnaiz JA, Castro A, Cosin J, Lekuona I, Guijarro C. Use of the cardiovascular polypill 40mg in secondary cardiovascular prevention. Clin Investig Arterioscler. 2018 Sep-Oct;30(5):240-247. doi: 10.1016/j.arteri.2018.04.004. Epub 2018 Jul 17. English, Spanish. PMID 30017176